CLINICAL TRIAL: NCT04649970
Title: Antegrade Double-J Stent Placement for the Treatment of Malignant Obstructive Uropathy: a Single Center Experience
Brief Title: Antegrade Double-J Stent Placement for the Treatment of Malignant Obstructive Uropathy
Status: Completed | Type: Observational
Sponsor: Université de Sousse (Other)
Responsible Party: Principal Investigator, ammar houssem, clinical professor, Université de Sousse
Other Study IDs: U23459
Record Dates: First submitted 2020-11-24; First posted 2020-12-02 (Actual); Last update posted 2020-12-04 (Actual); Status verified 2020-12

CONDITIONS: Urologic Neoplasms
MeSH Terms: conditions — Urologic Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- malignant uropathy: Antegrade double-J stent
  Interventions: Procedure: Antegrade double-J stent

INTERVENTIONS:
Procedure: Antegrade double-J stent — After exchanging the nephrostomy catheter over the J-tipped guidewire, 5 F multipurpose (45° tip) diagnostic vascular catheter was inserted. Once the pelvi¬ureteric junction was crossed and the ureter accessed, a straight hydrophilic guidewire and a catheter were used. Then, the cath-eter was advanced into the bladder over the wire, this guidewire was exchanged for an ultra-stiff guidewire, an 8 or 10 F double J ureteral stent was placed over the guidewire, and the safety kit of the stent was removed. A final fluoroscopic image was stored for correcting the stent position.

SUMMARY:
Ureteral double- J stent is usually inserted by retrograde approach for the treatment of obstructed upper urinary tract. The antegrade approach, can a suitable alternative in certain situations without the need for general or spinal anesthesia. The present study demonstrates the indications, success rate, and complications of this approach in the treatment of malignant obstructive uropathy.

DETAILED DESCRIPTION:
Data of consecutive patients in whom antegrade ureteral stent¬ing was performed between January 2013 and February 2020 were retrospectively analysed using patient records and radiology reports. A total of 174 patients (sexe ratio = 0.51, age range 9-91 years; mean age, 54 years) were included in the study.

Ureteral obstruction was caused by bladder cancer (n=92), uterin cancer (n=31), prostate cancer (n=28), colorectal cancer (n= 15) and retroperitoneal tumor (n= 8) (Table 1).

ELIGIBILITY:
Inclusion Criteria:

* malignant uropathy obstruction

Exclusion Criteria:

* benign uropathy obstruction

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: A total of 174 patients (sexe ratio = 0.51, age range 9-91 years; mean age, 54 years) were included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 174 (Actual)
Dates: Start 2013-01-01 (Actual); Primary Completion 2017-06-29 (Actual); Study Completion 2020-02-02 (Actual)

PRIMARY OUTCOMES:
number of patient having Antegrade double-J stent placement for the treatment of malignant obstructive uropathy | 7 years
  double j stent placement succeed or failed

CONTACTS AND LOCATIONS:
Overall Officials: ghaassen tlili, PROFESSOR, Study Director — university of sousse

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Tlili G, Ammar H, Dziri S, Ben Ahmed K, Farhat W, Arem S, Acacha E, Gupta R, Rguez A, Jaidane M. Antegrade double-J stent placement for the treatment of malignant obstructive uropathy: A retrospective cohort study. Ann Med Surg (Lond). 2021 Aug 16;69:102726. doi: 10.1016/j.amsu.2021.102726. eCollection 2021 Sep. PMID 34466220